CLINICAL TRIAL: NCT04146220
Title: Efficacy of Lower Dose Prednisolone in the Induction of Remission of Lupus Nephritis
Acronym: LN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Iftekhar Hussain Bandhan, Principal Investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSMMU/2018/8050
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Prednisolone; prednylidene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dose group (Experimental): Prednisolone 0.5 mg/kg/day
  Interventions: Drug: Prednisolone
- High dose group (Active Comparator): Prednisolone 1 mg/kg/day
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Prednisolone — Patients of the low and the high dose groups recieved prednisolone in different dose for initial 4 weeks, then tapered gradually. Both groups received pulse I/V methylprednisolone 500 mg/day daily for initial 3 days and monthly cyclophosphamide infusion 750-1000 mg/m2 body surface area.
  Other Names: Pred

SUMMARY:
The LN is a common cause of mortality and morbidity in SLE. The use of high-dose glucocorticoids (GC) with an immunosuppressive agent is usual practice for treating this condition. Higher dose of GC use might cause adverse effects along with clinical improvement. Studies had reported comparable outcome of lower dose of GC with minimum side effects. The aim of this study was to determine the outcome of lower dose prednisolone in the induction of remission of proliferative LN.

This prospective, clinical trial was conducted in Rheumatology outpatient and inpatient department of BSMMU from July 2018 to September 2019. Thirty-two subjects were enrolled after having informed consent. The ACR (American College of Rheumatology) criteria was followed for diagnosis of SLE. The patients of both genders, age ≥18 years, who fulfilled the ACR criteria of LN and unable to afford MMF were enrolled.

The patient evaluation tool was SELENA-DAI and Bengali version of SF-12 questionnaire. The 24-hour urinary protein, urine R/M/E, serum creatinine, CBC, serum C3, C4 levels and anti-dsDNA were done at baseline and at final visit of the study.

All patients received pulse I/V methylprednisolone 500 mg/day daily for 3 doses. After then experimental group received oral prednisolone 0.5 mg/kg/day and control group received oral prednisolone 1 mg/kg/day for a period of 4 weeks. After then the prednisolone was tapered by 10 mg/day in every two weeks until 40 mg/day, then 5 mg/day in every two weeks until 10 mg/day is reached, after two weeks the dose was tapered by 2.5 mg/day to a maintenance dose of 7.5 mg/day. Both groups were treated in the background of hydroxychloroquine (HCQ), angiotensin receptor blocker (ARB) and pulse I/V cyclophosphamide (CYC) for 6 cycle.

The ethical clearance was obtained from Institutional Review Board (IRB) of BSMMU and technical clearance was taken from rheumatology technical board.

DETAILED DESCRIPTION:
Rationale:

Lupus nephritis (LN) is a very common complication of systemic lupus erythematosus (SLE). Currently available all guidelines suggest an induction phase with glucocorticoids along with another immunosuppressive agent. However, the basis of using high dose of glucocorticoids are mostly empirical. There is no published data comparing low and high dose glucocorticoids in the treatment of LN. Use of high dose of glucocorticoids may increase morbidity like osteopenia, osteonecrosis of neck of femur, Cushing syndrome etc. Moreover, rate of infectious disease is very high in the investigator's country. Patient treated with high dose glucocorticoids may prone to develop serious infectious conditions. Researchers are currently trying to develop new regimen, which can replace the use of long-term glucocorticoids to treat LN. Unless the alternative regimen developed, well-controlled study is necessary to establish a lowest possible dose of glucocorticoid to treat this condition.

Research question:

Is lower dose prednisolone similar efficacious as the higher dose regimen in achieving complete remission of proliferative lupus nephritis?

Null hypothesis:

Lower dose prednisolone regimen is inferior to the higher dose regimen by more than - Δ in achieving the complete remission of proliferative lupus nephritis.

H0: P1-P2 ≤ - Δ P1 = Test drug (Prednisolone 0.5 mg/kg/day) P2 = Control drug (Prednisolone 1 mg/kg/day) Δ = Non-inferiority margin

Alternative hypothesis:

Lower dose prednisolone regimen is inferior to the higher dose regimen by less than - Δ in achieving the complete remission of proliferative lupus nephritis.

H1: P1-P2 > - Δ

General objective:

To assess efficacy of prednisolone 0.5 mg/kg/day in achieving remission of proliferative LN compared to 1 mg/kg/day

Specific objectives:

To compare:

* Changes of UTP level from the baseline to 24 weeks
* Changes of active urinary sediments level from the baseline to 24 weeks
* Changes of serum creatinine level from the baseline to 24 weeks
* Changes of quality of life from the baseline to 24 weeks
* Adverse effects during study period

Primary endpoint: (Time frame: at the end of 24th week)

• Complete renal remission

Secondary endpoints: (Time frame: at the end of 24th week)

* Renal remission (complete/partial) at 24 weeks
* Changes of UTP level from the baseline at 24 weeks
* Proportion of subjects with active urinary sediment at 24 weeks
* Changes of serum creatinine level from the baseline at 24 weeks
* Changes of eGFR from the baseline at 24 weeks
* Changes of anti-dsDNA level from the baseline at 24 weeks
* Changes of complements (C3 and C4) level from the baseline at 24 weeks
* Changes of SELENA-SLEDAI score from the baseline at 24 weeks
* Changes of SF-12 score from the baseline at 24 weeks

Study procedure:

This open labeled randomized controlled clinical trial was conducted in the outpatient and the inpatient department of Rheumatology, BSMMU from July 2018 to September 2019. Patients of SLE were interviewed after taking verbal consent. They were screened with history, physical examination, urine RME, 24hours UTP reports. Patients fulfilling the inclusion and exclusion criteria were enrolled in the study after taking informed written consent. Total 32 patients of SLE with proliferative LN were enrolled in the study. After the enrollment study subjects were randomized into experimental group (low dose group) and control group (high dose group) by lottery. Baseline laboratory tests were urine R/M/E, 24 hours UTP, serum creatinine, anti-dsDNA, C3, C4, CBC with ESR, SGPT. Baseline quality of life was assessed by Bengali version SF-12 questionnaire.

Both groups received pulse I/V methylprednisolone 500 mg/day daily for 3 doses. Then, patients of the low dose group received oral prednisolone 0.5 mg/kg/day (maximum 30 mg/day) and high dose group received oral prednisolone 1 mg/kg/day (maximum 60 mg/day) for initial 4 weeks. In the low dose group, prednisolone was tapered by 5 mg/day in every two weeks until 10 mg/day was reached, then after two weeks the dose was tapered by 2.5 mg/day to a maintenance dose of 7.5 mg/day. In the high dose group, prednisolone was tapered by 10 mg/day in every two weeks until 40 mg, then 5 mg/day in every two weeks until 10 mg/day is reached, after two weeks it was tapered by 2.5 mg/day to a maintenance dose of 7.5 mg/day.

Patients of both groups were treated with monthly CYC infusion, first dose 750 mg/m2 body surface area, subsequent doses were adjusted based on leukocyte nadir (≥ 4000 cells/mm3, doses were increased by 25%, to a maximum of 1 gm/m2 body surface area, the dose were reduced by 25% for leukocyte counts <4000 cells/mm3). Both groups of patients received hydroxychloroquine (HCQ), angiotensin receptor blocker (ARB) and other relevant medications. Patient education, vaccinations against influenza and pneumococcus were given to all the enrolled subjects. All patients were given Pneumocystis jirovecii prophylaxes.

Primary endpoint (complete remission) was assessed at the end of 24th week. Urine R/M/E, CBC with ESR, SGPT and serum creatinine were done in every 4 weeks. Twenty-four hours UTP were done at the end of 12 weeks and 24 weeks. Anti-dsDNA, C3 and C4 were done at the end of 24 weeks. Data were collected from a set of written questionnaires which was supplied to the patients and from physical examination and investigation findings. Quality of life was assessed by Bengali version of SF-12 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years of both sexes
2. Diagnosed case of systemic lupus erythematosus (SLE) as per ACR criteria
3. Patients consenting to participate in the study
4. Class III/IV lupus nephritis (LN) as evidenced by:

   * Confirmed proteinuria ≥ 500 mg/24 hours when assessed by 24-hour urine collection And
   * High titer anti-dsDNA (>75 U/ml) and low C3 (<0.9 g/l) and/or C4 (<0.1 g/l) Or
   * Kidney biopsy: with a histologic diagnosis of class III or IV lupus nephritis (International Society of Nephrology/Renal Pathology Society 2003 classification of lupus nephritis)

Exclusion Criteria:

1. Subjects not giving written informed consent
2. Pregnant or lactating women
3. Patient willing to be treated with MMF rather than CYC
4. Had taken CYC within 4 weeks prior to screening
5. Had taken >15 mg/day of prednisolone (or equivalent) for a period of >10 days during the previous month
6. Renal thrombotic microangiopathy
7. Estimated glomerular filtration rate (eGFR) as calculated by the Chronic Kidney Disease Epidemiology Collaboration equation of ≤45 mL/min/1.73 m2 at screening
8. Dialysis dependent patients, currently requiring renal dialysis (hemodialysis or peritoneal dialysis) or expected to require dialysis during the study period
9. A previous kidney transplant or planned transplant within study treatment period
10. Altered liver function (alanine aminotransferase greater than 2.5 times the upper limit of normal) at screening and confirmed before randomization
11. Malignancy
12. Lymphoproliferative disease or previous total lymphoid irradiation
13. Active bleeding disorders
14. Active tuberculosis (TB)
15. Diabetes mellitus
16. Any known hypersensitivity or contraindication to CYC, corticosteroids or any components of these drug products
17. Any overlapping autoimmune condition for which the condition or the treatment of the condition may affect the study assessments or outcomes (e.g., scleroderma with significant pulmonary hypertension; any condition for which additional immunosuppression is indicated)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Number of participants achieving complete renal remission | At the end of 24th week
  Complete renal remission is defined as a decline in the UTP level to <500 mg/day and return of serum creatinine to previous baseline.

SECONDARY OUTCOMES:
Number of participants achieving partial renal remission | At the end of 24th week
  Partial renal remission is defined as stabilization (±25%), or improvement of serum creatinine, but not to normal, and ≥50% decrease in UTP. If there was nephrotic-range proteinuria (UTP>3000 mg/day), improvement requires ≥50% reduction in UTP, and a UTP <3000 mg/day.

OTHER OUTCOMES:
Rate of achievement of normal anti-dsDNA level | At the end of 24th week
  A normal anti-dsDNA level is defined as anti-dsDNA <75 IU/ml
Rate of achievement of normal complements level | At the end of 24th week
  A normal complements level is defined as C3 <0.9 g/l and C4 <0.1 g/l
Rate of reduction of Safety of Estrogens in Systemic Lupus Erythematosus National Assessment - Systemic Lupus Erythematosus Disease Activity Index score | At the end of 24th week
  The Safety of Estrogens in Systemic Lupus Erythematosus National Assessment - Systemic Lupus Erythematosus Disease Activity Index (SELENA-SLEDAI) score ranges from 0 to 105. A higher score is associated with worse outcome. In clinical practice, a score ≤ 3 indicates "no flare", 3-12 indicates "mild to moderate flare", >12 indicates "severe flare".
Rate of improvement of Short Form-12 score | At the end of 24th week
  The Short Form-12 (SF-12) score includes the physical score (PCS-12) and the mental score (MCS-12). Both the PCS-12 and MCS-12 scores range from 0 to 100. A higher score is associated with better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Nazrul Islam, FCPS, MD, Study Chair — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hahn BH, McMahon MA, Wilkinson A, Wallace WD, Daikh DI, Fitzgerald JD, Karpouzas GA, Merrill JT, Wallace DJ, Yazdany J, Ramsey-Goldman R, Singh K, Khalighi M, Choi SI, Gogia M, Kafaja S, Kamgar M, Lau C, Martin WJ, Parikh S, Peng J, Rastogi A, Chen W, Grossman JM; American College of Rheumatology. American College of Rheumatology guidelines for screening, treatment, and management of lupus nephritis. Arthritis Care Res (Hoboken). 2012 Jun;64(6):797-808. doi: 10.1002/acr.21664. No abstract available. PMID 22556106
- [Background] Almaani S, Meara A, Rovin BH. Update on Lupus Nephritis. Clin J Am Soc Nephrol. 2017 May 8;12(5):825-835. doi: 10.2215/CJN.05780616. Epub 2016 Nov 7. PMID 27821390
- [Background] Bertsias GK, Tektonidou M, Amoura Z, Aringer M, Bajema I, Berden JH, Boletis J, Cervera R, Dorner T, Doria A, Ferrario F, Floege J, Houssiau FA, Ioannidis JP, Isenberg DA, Kallenberg CG, Lightstone L, Marks SD, Martini A, Moroni G, Neumann I, Praga M, Schneider M, Starra A, Tesar V, Vasconcelos C, van Vollenhoven RF, Zakharova H, Haubitz M, Gordon C, Jayne D, Boumpas DT; European League Against Rheumatism and European Renal Association-European Dialysis and Transplant Association. Joint European League Against Rheumatism and European Renal Association-European Dialysis and Transplant Association (EULAR/ERA-EDTA) recommendations for the management of adult and paediatric lupus nephritis. Ann Rheum Dis. 2012 Nov;71(11):1771-82. doi: 10.1136/annrheumdis-2012-201940. Epub 2012 Jul 31. PMID 22851469
- [Background] Buttgereit F, Straub RH, Wehling M, Burmester GR. Glucocorticoids in the treatment of rheumatic diseases: an update on the mechanisms of action. Arthritis Rheum. 2004 Nov;50(11):3408-17. doi: 10.1002/art.20583. No abstract available. PMID 15529366
- [Background] Seguro LP, Rosario C, Shoenfeld Y. Long-term complications of past glucocorticoid use. Autoimmun Rev. 2013 Mar;12(5):629-32. doi: 10.1016/j.autrev.2012.12.002. Epub 2012 Dec 20. PMID 23261815
- [Background] Ruiz-Irastorza G, Danza A, Perales I, Villar I, Garcia M, Delgado S, Khamashta M. Prednisone in lupus nephritis: how much is enough? Autoimmun Rev. 2014 Feb;13(2):206-14. doi: 10.1016/j.autrev.2013.10.013. Epub 2013 Nov 2. PMID 24189280
- [Background] Badsha H, Edwards CJ. Intravenous pulses of methylprednisolone for systemic lupus erythematosus. Semin Arthritis Rheum. 2003 Jun;32(6):370-7. doi: 10.1053/sarh.2002.50003. PMID 12833245
- [Background] Ruiz-Irastorza G, Danza A, Khamashta M. Glucocorticoid use and abuse in SLE. Rheumatology (Oxford). 2012 Jul;51(7):1145-53. doi: 10.1093/rheumatology/ker410. Epub 2012 Jan 23. PMID 22271756
- [Result] Austin HA 3rd, Klippel JH, Balow JE, le Riche NG, Steinberg AD, Plotz PH, Decker JL. Therapy of lupus nephritis. Controlled trial of prednisone and cytotoxic drugs. N Engl J Med. 1986 Mar 6;314(10):614-9. doi: 10.1056/NEJM198603063141004. PMID 3511372
- [Result] Boumpas DT, Austin HA 3rd, Vaughn EM, Klippel JH, Steinberg AD, Yarboro CH, Balow JE. Controlled trial of pulse methylprednisolone versus two regimens of pulse cyclophosphamide in severe lupus nephritis. Lancet. 1992 Sep 26;340(8822):741-5. doi: 10.1016/0140-6736(92)92292-n. PMID 1356175
- [Result] Gourley MF, Austin HA 3rd, Scott D, Yarboro CH, Vaughan EM, Muir J, Boumpas DT, Klippel JH, Balow JE, Steinberg AD. Methylprednisolone and cyclophosphamide, alone or in combination, in patients with lupus nephritis. A randomized, controlled trial. Ann Intern Med. 1996 Oct 1;125(7):549-57. doi: 10.7326/0003-4819-125-7-199610010-00003. PMID 8815753
- [Result] Illei GG, Austin HA, Crane M, Collins L, Gourley MF, Yarboro CH, Vaughan EM, Kuroiwa T, Danning CL, Steinberg AD, Klippel JH, Balow JE, Boumpas DT. Combination therapy with pulse cyclophosphamide plus pulse methylprednisolone improves long-term renal outcome without adding toxicity in patients with lupus nephritis. Ann Intern Med. 2001 Aug 21;135(4):248-57. doi: 10.7326/0003-4819-135-4-200108210-00009. PMID 11511139
- [Result] Houssiau FA, Vasconcelos C, D'Cruz D, Sebastiani GD, Garrido Ed Ede R, Danieli MG, Abramovicz D, Blockmans D, Mathieu A, Direskeneli H, Galeazzi M, Gul A, Levy Y, Petera P, Popovic R, Petrovic R, Sinico RA, Cattaneo R, Font J, Depresseux G, Cosyns JP, Cervera R. Immunosuppressive therapy in lupus nephritis: the Euro-Lupus Nephritis Trial, a randomized trial of low-dose versus high-dose intravenous cyclophosphamide. Arthritis Rheum. 2002 Aug;46(8):2121-31. doi: 10.1002/art.10461. PMID 12209517
- [Result] Mehra S, Usdadiya JB, Jain VK, Misra DP, Negi VS. Comparing the efficacy of low-dose vs high-dose cyclophosphamide regimen as induction therapy in the treatment of proliferative lupus nephritis: a single center study. Rheumatol Int. 2018 Apr;38(4):557-568. doi: 10.1007/s00296-018-3995-3. Epub 2018 Feb 15. PMID 29450636
- [Result] Appel GB, Contreras G, Dooley MA, Ginzler EM, Isenberg D, Jayne D, Li LS, Mysler E, Sanchez-Guerrero J, Solomons N, Wofsy D; Aspreva Lupus Management Study Group. Mycophenolate mofetil versus cyclophosphamide for induction treatment of lupus nephritis. J Am Soc Nephrol. 2009 May;20(5):1103-12. doi: 10.1681/ASN.2008101028. Epub 2009 Apr 15. PMID 19369404
- [Result] Sahay M, Saivani Y, Ismal K, Vali PS. Mycophenolate versus Cyclophosphamide for Lupus Nephritis. Indian J Nephrol. 2018 Jan-Feb;28(1):35-40. doi: 10.4103/ijn.IJN_2_16. PMID 29515299